CLINICAL TRIAL: NCT04453735
Title: MUscle Side-Effects of Atorvastatin in Coronary Patients (MUSE) -Follow-up Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vestre Viken Hospital Trust (Other)
Collaborators: The Hospital of Vestfold (Other); Oslo University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: REK 54041
Record Dates: First submitted 2020-06-28; First posted 2020-07-01 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2020-06

CONDITIONS: Statin Adverse Reaction
MeSH Terms: interventions — Tablets

STUDY DESIGN:
Intervention Model Description: Prospective, open, intervention study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Atorvastatin mylan 40 mg once daily
  Interventions: Drug: Atorvastatin mylan 40 Mg Oral Tablet
- Control (No Intervention): No statin therapy

INTERVENTIONS:
Drug: Atorvastatin mylan 40 Mg Oral Tablet — Oral tablet on regular prescription
  Arms: Intervention

SUMMARY:
Statins are cornerstone treatment in secondary cardiovascular disease (CVD) prevention. Today, statin non-adherence (patients not taking their prescribed drug) remains a major public health concern, leading to adverse outcomes in terms of morbidity, mortality and healthcare costs. The principal reason for statin non-adherence and discontinuation is statin-associated muscle symptoms (SAMS). Objective SAMS diagnostics do not exist. We aim to unravel the pathophysiology of SAMS and develop diagnostic tools to differentiate real SAMS from muscle symptoms not related to the statin, among coronary patients with self-perceived SAMS. In this follow-up study we aims to determine the effect of 7 weeks open treatment with atorvastatin 40 mg/day, followed by 7 weeks open treatment with no lipid lowering treatment, on muscle symptom intensity in patients classified with confirmed statin-associated muscle symptoms (SAMS) (i.e. statin-dependent muscle side-effects) and non-SAMS in the MUscle Side-Effects of atorvastatin in coronary patients (MUSE) randomized double blinded cross-over trial.

We have developed novel methods that will be used to measure atorvastatin metabolites and drug effect biomarkers directly in skeletal muscle and blood . The diagnostic accuracy of these biomarkers to differentiate real SAMS from non-SAMS will be evaluated. A new diagnostic tool may potentially be implemented to assess SAMS in the individual patient and enable personalized follow-up. It may also represent an important tool in the communication with patients misattributing their muscle symptoms to statins. The long-term results may be better quality of life and reduced morbidity, mortality and healthcare costs.

ELIGIBILITY:
Inclusion Criteria:

* Participation in the MUSE trial (Eudract nr. 2018-004261-14) and still fulfilling the study entry criteria: First or recurrent diagnosis (myocardial infarction) or treatments (PCI or CABG) for a CHD event 12-42 months prior to study start.

Exclusion Criteria:

* First or recurrent diagnosis (myocardial infarction) or treatments (PCI or CABG) for a CHD event the a) past 12 months prior to study start in high risk patients (i.e. at least one of following comorbid conditions: systolic heart failure, >1 previous myocardial infarction, kidney failure, diabetes, and smokers) and b) the past 6 months prior to study start in low risk patients without any of the co-morbid conditions mentioned above and in patients who are not taking a statin at all.
* Patients with symptomatic peripheral artery disease and patients with familial hypercholesterolemia
* Patient has any contraindications for atorvastatin listed in the Summary of Product Characteristics (i.e. known hypersensitivity to the ingredients, acute liver failure/ ALT > 3 times upper limit of the normal range in blood at study start, pregnancy and breastfeeding )
* History of previous rhabdomyolysis, myopathy or liver failure due to statin treatment with CK > 10 times upper limit of the normal range or ALT > 3 times upper limit of the normal range.
* Any condition (e.g. psychiatric illness, dementia) or situation, that in the investigator's opinion could put the subject at significant risk, confound the study results, interfere significantly with the subject participation in the study, or rendering informed consent unfeasible
* Short life expectancy (<12 months) due to other medical conditions
* Not being able to understand Norwegian.
* Women of childbearing potential defined as all premenopausal female.
* Participation in another randomized clinical trial
* Classified with significantly more muscle symptoms on placebo than on atorvastatin in the MUSE trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2020-08-19 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2020-12-18 (Actual)

PRIMARY OUTCOMES:
Individual mean difference in muscular symptom intensity measured with a 0 (no symptoms) to 10 (worst imaginable symptoms) Visual Analogue Scale (VAS) score between treatment periods with statin and "no statin treatment" | 16 weeks following study start
  Individual mean difference in muscular symptom (i.e. pain, aching, tenderness, stiffness, cramp and/or weakness) intensity between treatment periods with statin and no statin, reported by the patients over the last three weeks (i.e. week 4-7) measured with a 0 (no symptoms) to 10 (worst imaginable symptoms) Visual Analogue Scale (VAS) score with aggregated data from each subscale

SECONDARY OUTCOMES:
The proportion of patients who report muscle symptoms on atorvastatin treatment and not on statin (dichotomous Statin Associated Muscle Symptom classification) | 16 weeks following study start
Correlation between atorvastatin-related variables in muscle and the primary study endpoint. The ability of atorvastatin-related variables in muscle to differentiate confirmed SAMS and non-SAMS | 16 weeks following study start
Correlation between atorvastatin-related variables in plasma vs. muscle and PBMC vs. muscle. Correlation between atorvastatin-related variables in blood and the primary study endpoint. | 16 weeks following study start
Correlation between atorvastatin: HMGCR in muscle and the primary study endpoint. The ability of atorvastatin:HMGCR in muscle to differentiate confirmed SAMS and non-SAMS. | 16 weeks following study start
Correlation between atorvastatin:HMGCR in PBMC vs. muscle. Correlation between atorvastatin:HMGCR in PBMC and the primary study endpoint. | 16 weeks following study start
Correlation between mevalonate pathway intermediates in muscle and the primary study endpoint. The ability of mevalonate pathway intermediates in muscle to differentiate confirmed SAMS and non-SAMS. | 16 weeks following study start
Correlation between mevalonate pathway intermediates in plasma vs. muscle and PBMC vs. muscle. Correlation between mevalonate pathway intermediates in blood and the primary study endpoint. | 16 weeks following study start
Correlation between mitochondrial respiratory enzymes in muscle and the primary study endpoint. The ability of mitochondrial respiratory enzymes in muscle to differentiate confirmed SAMS and non-SAMS. | 16 weeks following study start
Correlation between mitochondrial respiratory enzymes in PBMC vs. muscle. Correlation between mitochondrial respiratory enzymes in PMBC and the primary study endpoint. | 16 weeks following study start
Correlation between the FKBP1A:RyR1 ratio in muscle and the primary study endpoint. The ability of the FKBP1A:RyR1 ratio in muscle to differentiate confirmed SAMS and non-SAMS. | 16 weeks following study start
Correlation between the FKBP1A:RyR1 ratio in PBMC vs. muscle. Correlation between the FKBP1A:RyR1 ratio in PBMC and the primary study endpoint. | 16 weeks following study start
Correlation between caspase 3 signalling in muscle and the primary study endpoint. The ability of caspase 3 signalling in muscle to differentiate confirmed SAMS and non-SAMS. | 16 weeks following study start
Correlation between caspase 3 signalling in PBMC vs. muscle. Correlation between caspase 3 signalling in blood and the primary study endpoint. | 16 weeks following study start
Difference in muscle response variables between atorvastatin period and non-statin period. | 16 weeks following study start
Correlation of molecular effects in blood vs. muscle. Difference in blood response variables between atorvastatin period and non-statin period. Correlation between atorvastatin-related variables and response variables in blood. | 16 weeks following study start
Statin adherence measured with indirect methods and by parent drug and metabolite concentrations in blood | 16 weeks following study start
New-onset CHD symptoms. Intolerable muscle symptoms leading to discontinuation from the treatment arm. Creatine kinase (CK) > 10 times upper limit of the normal range or alaninaminotransferase (ALT) > 3 times upper normal limit | 16 weeks following study start

CONTACTS AND LOCATIONS:
Locations (2):
- Norway (2):
  - Vestre Viken HF, Drammen Hospital, Drammen, Buskerud
  - Hospital of Vestfold, Tønsberg, Vestfold

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be made available for other researchers
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available within 5 years of study completion